CLINICAL TRIAL: NCT05104112
Title: Evaluation of a Therapeutic Education Program for Pregnant Women with a First Child Diagnosed with an Autism Spectrum Disorder (ASD)
Brief Title: Evaluation of a Therapeutic Education Program for Pregnant Women with a First Child Diagnosed with an Autism Spectrum Disorder
Acronym: AUTMER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP191096
Record Dates: First submitted 2021-10-11; First posted 2021-11-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Child Psychiatry
Keywords: autism spectrum disorder; therapeutic education; prevention; pregnancy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: A pragmatic, multicenter, randomized, delayed-onset, stepped-wedge cluster study.
Who Masked: Outcomes Assessor
Masking Description: To ensure blinding, the primary endpoint, assessed on video, will be measured at the end of the study by a blinded investigator from the randomization group and from a different center than the inclusion center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Pregnant women followed by the center in the period before the intervention is implemented (the start of which is determined by randomization)
- experimental group (Experimental): Pregnant women followed by the center during the period after the intervention is implemented (the start of which is determined by randomization)
  Interventions: Other: The M.E.R. program

INTERVENTIONS:
Other: The M.E.R. program — The M.E.R program is a therapeutic education intervention for mothers of children with ASD during a new pregnancy. This program, which is a pilot in France and in Europe, involves several dimensions, both pedagogical and behavioral (strategies for stimulating the baby, use of specific communication and interaction tools) and psychological (reduction of stress, anxiety, etc. in the mother).
  It includes 8 individual interviews of 1h30 every 15 days. The first and the last one are for evaluation purposes, the 6 intermediate sessions constitute the accompaniment. The structure of the program and the sessions are based on what is recommended in therapeutic education. The sessions can take place on the hospital site or at home.
  Arms: experimental group

SUMMARY:
Autism Spectrum Disorder (ASD) is a heterogeneous set of severe developmental abnormalities of the nervous system characterized by deficits affecting social interactions and verbal and non-verbal communication, as well as the presence of restricted interests, repetitive behaviors, and atypical sensory manifestations . ASD affects approximately 1% of the general population (Elsabbagh et al., 2012). Studies of siblings of individuals with ASD show that ASD is present in 7-20% of the offspring in families where a child has had a diagnosis of ASD and this prevalence increases if there are two diagnosed children.

Several studies show the benefits of interventions targeting parents' interaction strategies in the early phases of development of infants at high risk for ASDs, in reducing the risk itself or its severity. Very early intervention, due to the presence of significant brain plasticity at these stages, may be particularly effective in changing these emerging trajectories, from a "preventive intervention" perspective that would aim to mitigate developmental risk and alter prodromal symptom trajectories, rather than eliminate a condition.

Our hypothesis is that the implementation of a specific therapeutic education program during a new pregnancy in the mother of a child with a diagnosis of ASD (MER Program) could improve the mother's well-being, increase parenting communication skills, and thereby improve interaction with the newborn at high risk for ASD. If the infant is affected, it may also reduce the symptoms of the disorder. Indirectly, it could also improve the well-being of the other parent involved in the interaction.

The M.E.R (Mères Ecoute Ressources) programme is a therapeutic education intervention aimed at mothers of children with ASD during a new pregnancy. This programme, which is being piloted in France and Europe, involves a number of dimensions, both educational and behavioural (strategies for stimulating the baby, use of specific communication and interaction tools) and psychological (reduction of stress, anxiety, etc. in the mother).

The programme comprises 8 one-to-one sessions lasting 1.5 hours every 15 days. The first and last of these are for assessment purposes, with the 6 intermediate sessions constituting the support. The structure of the programme and the sessions is based on what is recommended in therapeutic education. The sessions can take place on the hospital site or by teleconsultation (remote consultation used in the context of healthcare).

DETAILED DESCRIPTION:
Randomized controlled trial with deferred start, French multicenter stepped-wedge type.

The start date of the intervention in each center will be done by randomization, defining 2 periods: a control period located before the start of the intervention, and an experimental period located after the start of the intervention.

This design allows the principal investigating team to train the centers associated in turn with the intervention, and to have a control group with structured follow-up but without intervention.

All subjects will be included before 26 ADT and assigned to the control or experimental group, depending on the time of inclusion and the randomization of the center to which they belong.

The follow-up will be conducted in 2 phases: 1. during pregnancy and 2. After the birth of the child.

Subjects included were pregnant women who already had a child with an ASD diagnosis, the second parent if present, and the newborn at risk for an ASD diagnosis.

The primary objective of this study is to evaluate the effect of an innovative therapeutic education program (the MER program) versus control in pregnant women with a first child followed for ASD on the quality of interaction strategies of the mother-infant dyad at 10 months postpartum.

The primary endpoint was the caregiver non-directiveness subscore of the Manchester Assessment of Caregiver-infant Interaction (MACI) scale at 10 months postpartum. This subscore is both the most sensitive to intervention and predictive of ASD diagnosis.

The first secondary objective is the evaluation of the effect of the MER versus control program on:

* maternal pregnancy-related anxiety (PRAQ-R2 score) ;
* Anxious and depressive symptomatology and quality of life (WhoQoL-Bref score) in the mother and the second parent during pregnancy (EPDS score) and up to 20 months of age of the newborn (HAM-Anxiety and HAM-Depression scores);
* perceived stress related to pregnancy (ALES score)
* mother-infant interaction at 10 and 20 months (MACI score and subscore);
* autistic signs in at-risk infants at 20 months (ADOS Toddler score);

The second secondary objective was to study variables that could impact the effect of the intervention, including

* adherence: compliance with sessions, satisfaction of participants (PEI-Parent score) ;
* other variables that could modulate the effect of the intervention: sociodemographic variables (socioeconomic level, family configuration, number of children); clinical profile of the mother (intellectual efficiency (Raven's PM score), psychiatric comorbidities (DIGS, SRS score)); clinical profile of the child already diagnosed (ADI-R and ADOS score; developmental level); clinical profile of the infant at risk (gestational age, MSEL, IBQ-R and ECBQ scores).

The third secondary objective was to describe the barriers and levers to the implementation of the intervention.

Characteristics related to the implementation of the intervention (recruitment, uptake, fidelity, and implementation) will be collected, as well as the profile of mothers who did not participate in the project.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of children with a diagnosis of ASD, in pregnancy (before the 26th week of amenorrhea);
* The diagnosis of ASD of the older child has been made, according to the DSM IV-TR or DSM 5 criteria, formalized by a diagnostic evaluation including: the Autism Diagnostic Observation Schedule ADOS, the Autism Diagnostic Interview - Revised version (ADI-R) accompanied by a cognitive evaluation of the child (Wechsler/Mullen Scales of Early Learning/Raven's Progressive Matrices);
* Informed consent from mother and sec

Exclusion Criteria:

* Presence of a clearly identified and unstabilized severe psychiatric disorder in the mother (confirmed by medical interview and DIGS questionnaire conducted at the time of the inclusion visit) and/or intellectual disability;
* Engagement in another form of individual therapeutic intervention.
* Refusal of either parent (for child assessment, primary criterion)
* Parents not proficient in French language
* Persons (mother or second parent) under legal protection, guardianship or trusteeship, persons deprived of liberty, under court protection, under psychiatric care, under constraint, admitted to a health or social institution for purposes other than research
* Persons with cognitive disorders or intellectual disabilities

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Manchester Assessment of Caregiver-infant Interaction (MACI) "caregiver non-directiveness" subscore | 5 months after delivery
  mother-baby interaction in the experimental group versus the control group at 5 months postpartum.
  This subscore is the most sensitive to intervention and predictive of ASD diagnosis.

SECONDARY OUTCOMES:
Pregnancy-Related Anxiety Questionnaire-Revised2 (PRAQ-R2) subscore | between 11 weeks and 26 weeks of gestation
  To evaluate the effect of the MER program on maternal anxiety related to pregnancy
Pregnancy-Related Anxiety Questionnaire-Revised2 (PRAQ-R2) subscore | at 3 months after intervention
  To evaluate the effect of the MER program on maternal anxiety related to pregnancy
Appraisal of Life Events Scale (ALES) | between 11 weeks and 26 weeks of gestation
  Perceived pregnancy-related stress in the mother.scale with a list of adjectives, rated on a five-point Likert scale)
Appraisal of Life Events Scale (ALES) | at 3 months after intervention
  Perceived pregnancy-related stress in the mother.scale with a list of adjectives, rated on a five-point Likert scale
Edimburgh Postnatal Depression Scale (EPDS) | 10 months after birth
  used to assess the risk of postnatal depression and is useful for identifying the presence of anxiety symptoms.The threshold retained for the French validation is 10.5, above which a depression is possible and below which the risk is very low.
quality of life score-Bref (WhoQol-Bref) | 10 months after birth
  WHOQOL-BREF includes 26 items that measure the following broad domains: physical health, psychological health, social relationships and environment.
parental anxiety score (HAM) | 10 months after birth
  hetero-questionnaire with 14 items, measuring both the psychic (mental agitation and psychological distress) and somatic (physical complaints related to anxiety) expression of anxiety. Each item is rated on a Likert scale from 0 to 4 (total range 0-56, where <17= mild anxiety; 18-24= mild to moderate; 25-30 moderate to severe)
mother's intelligence quotient | between 11 weeks and 26 weeks of gestation
  measured by Raven's Progressive Matrices
Social Responsiveness Scale (SRS) | between 11 weeks and 26 weeks of gestation
  to refine the evaluation of social difficulties in a dimensional way
Wechsler Mullen scale | between 11 weeks and 26 weeks of gestation
  developmental level of the ASD child

CONTACTS AND LOCATIONS:
Overall Officials: Anita Beggiato, PHD, Principal Investigator — APHP
Locations (1):
- Hôpital Robert Debré, Paris, Paris, France